CLINICAL TRIAL: NCT01464398
Title: Stress Reduction for PCOS and Non-PCOS Women
Brief Title: Stress Reduction for Overweight or Obese Women Either With Polycystic Ovary Syndrome (PCOS) or Without PCOS (Non-PCOS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Nazia Raja-Khan, M.D., Assistant Professor of Medicine, Division of Endocrinology, Diabetes, and Metabolism, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 34145EP; K23AT006340 (NIH)
Record Dates: First submitted 2011-10-31; First posted 2011-11-03 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Polycystic Ovary Syndrome; Overweight; Obesity; Stress, Physiological; Stress, Psychological
Keywords: Polycystic Ovary Syndrome; stress; mindfulness; meditation; health education; women; overweight; obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Overweight; Obesity; Stress, Psychological; Health Education | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stress reduction (Active Comparator): Mindfulness-based stress reduction
  Interventions: Behavioral: Stress reduction
- Stress reduction with Health education (Active Comparator): General stress management and health education
  Interventions: Behavioral: Stress reduction with Health education

INTERVENTIONS:
Behavioral: Stress reduction — 8 weekly sessions
  Arms: Stress reduction
Behavioral: Stress reduction with Health education — 8 weekly sessions
  Arms: Stress reduction with Health education

SUMMARY:
The purpose of this study is to determine the effects of stress reduction on glucose, blood pressure, quality of life and overall health and well-being in overweight or obese women, either with Polycystic Ovary Syndrome (PCOS) or without PCOS (non-PCOS). Stress reduction treatment sessions will include one or more of the following activities: breathing exercises, meditation, stretching exercises or health education activities.

ELIGIBILITY:
Inclusion Criteria:

1. Women, age 18 years or older
2. Body mass index (BMI) ≥ 25 kg/m2 (overweight or obese)

Exclusion criteria:

1. Current pregnancy
2. Secondary causes of hyperandrogenemia, such as known or suspected androgen secreting tumors, Cushing's syndrome, or hyperprolactinemia (prolactin >30)
3. Untreated hypothyroidism or hyperthyroidism (defined as TSH <0.2 or >5.5 mIU/mL)
4. Severe active neuropsychological disorder such as psychosis or suicidal ideation
5. Severe untreated depression or anxiety. Women with severe depression or anxiety will be allowed to participate if they are under the care of a mental health specialist as long as they have permission to do so from their mental health specialist and will continue to follow-up with their mental health specialist during the study.
6. History of an inpatient admission for psychiatric disorder within the past two years
7. Active alcohol or drug abuse
8. Inability to read, speak or write English
9. Inability to commit to the intervention and follow-up
10. Current enrollment in a stress reduction program
11. Mindfulness practice within the past 6 months (regular formal practice at least once a week)
12. Current enrollment in other investigative studies
13. Type 1 diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Toronto Mindfulness Scale at 8 weeks | baseline and 8 weeks

SECONDARY OUTCOMES:
Change from Baseline in Toronto Mindfulness Scale at 16 weeks | baseline and 16 weeks
Change from Baseline in Hemoglobin A1c at 8 weeks | baseline and 8 weeks
Change from Baseline in Hemoglobin A1c at 16 weeks | baseline and 16 weeks
Change from Baseline in Mean Arterial Pressure at 8 weeks | baseline and 8 weeks
Change from Baseline in Mean Arterial Pressure at 16 weeks | baseline and 16 weeks
Change from Baseline in SF-36 at 8 weeks | baseline and 8 weeks
Change from Baseline in SF-36 at 16 weeks | baseline and 16 weeks
Change from Baseline in Brief Symptom Inventory-18 at 8 weeks | baseline and 8 weeks
Change from Baseline in Brief Symptom Inventory-18 at 16 weeks | baseline and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nazia Raja-Khan, MD, Principal Investigator — Pennsylvania State University College of Medicine
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Raja-Khan N, Agito K, Shah J, Stetter CM, Gustafson TS, Socolow H, Kunselman AR, Reibel DK, Legro RS. Mindfulness-Based Stress Reduction in Women with Overweight or Obesity: A Randomized Clinical Trial. Obesity (Silver Spring). 2017 Aug;25(8):1349-1359. doi: 10.1002/oby.21910. Epub 2017 Jul 7. PMID 28686006
- [Derived] Raja-Khan N, Agito K, Shah J, Stetter CM, Gustafson TS, Socolow H, Kunselman AR, Reibel DK, Legro RS. Mindfulness-based stress reduction for overweight/obese women with and without polycystic ovary syndrome: design and methods of a pilot randomized controlled trial. Contemp Clin Trials. 2015 Mar;41:287-97. doi: 10.1016/j.cct.2015.01.021. Epub 2015 Feb 7. PMID 25662105